CLINICAL TRIAL: NCT02613975
Title: A Cross Over Case Control Study Using a Vibration Positional Device for Treatment of Position Dependent Obstructive Sleep Apnea
Brief Title: A Cross Over Case Control Study of a Vibration Positional Device for Treatment of OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Doctor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2013.689
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: OSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- on positional device (Experimental): patients who could not tolerate cpap will be provided with positional device for treatment of OSA which will vibrate when patients lie in prone position
  Interventions: Device: positonal device
- patients on dental device (Experimental): patients on dental devices but not optimally treated for OSA will be provided positional device for optimization of treatment for OSA, which will vibrate when patients lie in prone position
  Interventions: Device: positonal device

INTERVENTIONS:
Device: positonal device — positional device detects prone positional and will vibrate to cause patient to lie laterally

SUMMARY:
Positional therapy is considered as a kind of conservative treatment especially for patients with OSA which varies with body positions, and has been reported to be useful in selected cases especially those with positional OSA. Positional OSA is present when the overall apnea hyponea index (AHI) is > 5/hr with a supine AHI being more than 2 times of AHI in other positions, in a symptomatic patient. There will be 2 groups of patients in this study. Group 1 consists of patients with positional OSA who refuse CPAP or tolerate CPAP poorly. They will be provided with a vibration device as treatment, which will be worn on the neck during sleep. This device senses the position of the patient during sleep. It will vibrate when the patient lies supine until the patient turns laterally, thus prevents the patient to lie flat during sleep and reduce the severity of OSA. It will be switched on and off for a period of 15 days alternatively with sleep study performed at the end of each period respectively to determine its efficacy in the on and off mode. There will be a wash out period of 1 week in between the on and off period to remove any residual effect. Group 2 consists of patients with positional OSA who are using dental device but response or tolerated poorly. They will use the vibration device with dental device together as dual therapy, to assess the role of combination therapy. The device will be operated in on and off mode with sleep study being performed in a similar manner as in group 1. Informed consent will be signed. Each participant will have 2 sleep studies performed at home, which will be supported technically by technician visiting their home for hook up of necessary equipment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with position dependent OSA which is defined as supine AHI >2 times the AHI in other positions, while an overall AHI >5/hr.
2. Patients who cannot tolerate/not using CPAP.
3. Patients who are on dental devices but residual AHI is > 15 and symptomatic.
4. Patients consent to study and able to follow the instruction of using positional device and home sleep study device.

Exclusion Criteria:

1. Patients with pregnancy.
2. Patients who refuse home sleep studies.
3. Patients with parasomnias.
4. Patients who cannot follow the instruction of using positional device or home sleep study device.
5. Patients who tolerate CPAP well with good treatment outcome.
6. Patients on dental device with good symptoms improvement and residual AHI < 15/hr

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Reduction of AHI using the positional device | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kin Wang To, MBChB, Principal Investigator — Honoary clinical assistant professor
Locations (1):
- Department of Medicine and Therapeutics, Prince of Wales Hospital, CUHK, Shatin, Hong Kong